CLINICAL TRIAL: NCT02911649
Title: Reducing Sedentary Behaviour Through Wearable Technology and Education
Brief Title: Reducing Sedentary Behaviour With Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-5437
Record Dates: First submitted 2016-08-08; First posted 2016-09-22 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Fatigue; Prostate Cancer; Breast Cancer; Sedentary Behaviour; Physical Activity
MeSH Terms: conditions — Fatigue; Prostatic Neoplasms; Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Wearable Device Only (Experimental): Participants will be allowed to choose one of three wearable devices (FitBit, Garmi or Polar), for the wearable technology intervention. Once the participant has chosen their wearable device they will be oriented to their chosen device, platform to obtain information from the device, as well as a guide with ideas for reducing sedentary behaviour. Participants will be asked to wear the devices every day during waking hours.
  Interventions: Other: Wearable Technology - Garmin Vivosmart; Other: Wearable Technology - FitBit Alta; Other: Wearable Technology - Polar Loop 2
- Online Educational Workshop Only (Experimental): The Online Educational Group will be asked to participate in 6 online workshops that will occur during the 12-week intervention. Adobe connect software will be used to implement these workshops which allows for interaction between participants and leader. Workshops will focus on specific aspects related to reducing sedentary behaviours and increasing PA time. Each workshop will be developed by study coordinator/author (MO) and constructed using Social Cognitive Theory (SCT), ensuring the themes such as self-efficacy, self-control and reinforcements are within each topic. EDU topics will include motivation, goal setting, and activities and ways to reduce sedentary behaviour.
  Interventions: Other: Online Educational Group
- Wearable Device+Online Edu Workshop (Experimental): Both the wearable technology intervention and Online Educational Group intervention simultaneously.
  Interventions: Other: Wearable Technology - Garmin Vivosmart; Other: Online Educational Group; Other: Wearable Technology - FitBit Alta; Other: Wearable Technology - Polar Loop 2
- Control Group (No Intervention): Participants in this group will receive usual care

INTERVENTIONS:
Other: Wearable Technology - Garmin Vivosmart — Wearable devices will be used to show participants their activity levels daily, as well as weekly overview of their activity levels.
  Arms: Wearable Device Only; Wearable Device+Online Edu Workshop
Other: Online Educational Group — A workshop leader will lead participants through an educational workshop and group discussion on topics related to reducing sedentary behaviour
  Arms: Online Educational Workshop Only; Wearable Device+Online Edu Workshop
Other: Wearable Technology - FitBit Alta — Wearable devices will be used to show participants their activity levels daily, as well as weekly overview of their activity levels.
  Arms: Wearable Device Only; Wearable Device+Online Edu Workshop
Other: Wearable Technology - Polar Loop 2 — Wearable devices will be used to show participants their activity levels daily, as well as weekly overview of their activity levels.
  Arms: Wearable Device Only; Wearable Device+Online Edu Workshop

SUMMARY:
Cancer-related fatigue (CRF) can be experienced by individuals with Prostate Cancer (PC), which can have profound effects on their well-being. Although physical activity has been shown to improve CRF, the recommended levels are generally not met. Step count and distance traveled information can help individuals to increase their physical activity. Wearable technology (WEAR) provides the user with feedback of their physical activity which can motivate behaviour change. Similarly, education workshops (EDU) on the effects of sedentary behaviour and physical activity may also reduce sedentary behaviour.

The objectives of this study are to evaluate the effects of WEAR and EDU on sedentary behaviour and CRF, and to explore the feasibility of WEAR in this population. Participants in this study will be randomly assigned into WEAR, EDU, WEAR+EDU, or control over a three-month intervention. Assessments at baseline, post-intervention and a 3-month follow up will evaluate CRF, quality of life and level of sedentary behaviour, and use of WEAR devices.

The results from this study will provide evidence-based knowledge on the impact of WEAR and EDU on sedentary behaviour and CRF, and an understanding on the use of technology within the PC population. These results can shape the development of programming for CRF and the use of scale-able technology-based interventions/approaches in this population.

ELIGIBILITY:
Inclusion Criteria:

* PC survivors aged 18 years or older
* Currently sedentary, defined as <90 minutes per week of activity
* Fluent in English
* Access to a computer with internet connectivity

Exclusion Criteria:

• Men who are or have received chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  At baseline we will evaluate the recruitment rate of participants for the feasibility of this trial and reasons for declining to participate
Retention rate | 3 month assessment (Post-Intervention)
  At the end of the intervention and follow-up assessment, we will measure retention rate through number of participants who have withdrawn from the study.
Adherence | 3 month assessment (Post-Intervention)
  Adherence will be measured for participants attendance throughout the intervention.
WEAR device preference | 3 month assessment (Post-Intervention)
  This will be measured through the number of participants that choose each of the three devices.
Acceptability | 6 months assessment (follow-up)
  Acceptability will be measured through the end of study questionnaire at the follow-up assessment
Outcome measures captured | 6 month assessment (follow-up)
  This will be measured through review and analysis of data obatined for completeness

SECONDARY OUTCOMES:
Cancer-Related Fatigue | Baseline, 3 month assessment(post-intervention), 6 month assessment (3 month Follow up)
  Assessed with Functional Assessment of Cancer Therapy - Fatigue (FACT-F)
Sedentary Behaviour | Baseline, 3 month assessment(post-intervention), 6 month assessment (3 month Follow up)
  Assessed through accelerometry and Sit-Q 7 Day questionnaire
Quality of Life | Baseline, 3 month assessment(post-intervention), 6 month assessment (3 month Follow up)
  Assessed with Functional Assessment of Cancer Therapy - General (FACT-G)
Depression | Baseline, 3 month assessment(post-intervention), 6 month assessment (3 month Follow up)
  Assessed with Patient Health Questionnaire - 9 (PHQ-9)
Understand attitudes towards using wearable technology | Baseline, 3 month assessment(post-intervention), 6 month assessment (3 month Follow up)
  Assessed through semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD MSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No